CLINICAL TRIAL: NCT01253148
Title: Phase II Study Of Intrahepatic Arterial Injection of 90-Y Glass Microspheres As First-Line Treatment For Cholangiocarcinoma
Brief Title: Study Of Intrahepatic Arterial Injection of 90-Y Glass Microspheres for Cholangiocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16236; NCI-2011-00794 (Other: NCI CTRP)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Cholangiocarcinoma
Keywords: Liver; Bile Duct
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Microspheres; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arterial Injection of 90-Y Microspheres (Experimental): Intrahepatic Arterial Injection of 90-Y Glass Microspheres as First-Line Treatment For Cholangiocarcinoma
  Interventions: Device: TheraSphere® Yttrium-90 (Y-90) Microspheres

INTERVENTIONS:
Device: TheraSphere® Yttrium-90 (Y-90) Microspheres — Y-90 is incorporated into very tiny glass beads called microspheres and is injected into the liver through the blood vessels supplying the liver.
  Other Names: 90y; Intrahepatic Arterial Injection; Radiotherapy; Radioactive Microspheres; Yttrium Glass Microspheres

SUMMARY:
The purpose of this study is to see if Therasphere will be a better way to treat cholangiocarcinoma. The investigators want to find out what effects, good and/or bad, this treatment will have on the patient and their cancer.

DETAILED DESCRIPTION:
The goal of treatment with TheraSphere is to allow a large dose of radiation to be delivered directly to the tumor with less risk of toxic effects from radiation to other parts of the body or to healthy liver tissue when compared with currently available treatments.

The standard treatment for cholangiocarcinoma is surgery (if possible), external beam radiation therapy and/or chemotherapy. External beam radiation therapy to the liver may reduce symptoms, but only 20% of patients experience significant tumor shrinkage. Chemotherapy has response rates ranging from 6-19%. More recently, a new approach has been developed, called TheraSphere. Based on the results of earlier studies with TheraSphere, the study doctors at Moffitt feel this is a reasonable alternative to the standard treatment for this disease.

TheraSphere has restricted approval from the United States Food and Drug Administration (FDA) for the treatment of hepatocellular liver cancer; but it has not yet been approved for the treatment of cholangiocarcinoma. TheraSphere is a medical device containing yttrium-90 (Y-90), a radioactive material that has been used previously in the treatment of liver tumors. Y-90 is incorporated into very tiny glass beads called microspheres and is injected into the liver through the blood vessels supplying the liver.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed or recurrent (post surgery) histologically or cytologically proven cholangiocarcinoma.
* Patients can have solitary, multifocal unilobar, or bilobar disease without evidence of extrahepatic involvement. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with spiral computed tomography (CT) scan or magnetic resonance imaging (MRI).
* Age >18 years
* Life expectancy of greater than 3 months based on physician judgment
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2 (Karnofsky 50%)
* No prior chemotherapy or radiation treatment for cholangiocarcinoma
* Childs-Pugh score A or Childs-Pugh score B without portal vein thrombus
* Lung shunting that predicts lung dose to be <30 Gy in a single treatment
* The effects of TheraSpheres on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because radioactive spheres are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document
* Adequate baseline hematopoietic function:

  * total white blood cell count equal to or greater than 3,000/mm³
  * absolute granulocyte count greater than 1,500/mm³
  * platelet count equal to or greater than 100,000/mm³
  * Hemoglobin >8.0

Exclusion Criteria:

* Patients receiving any other investigational agents
* Patients with extrahepatic disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because TheraSpheres are radioactive and radiation is a known agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TheraSpheres, breastfeeding should be discontinued if the mother is treated with TheraSpheres.
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. In addition, antiretrovirals are known radiation sensitizers and could dramatically increase the risk of fulminant hepatic failure. Therefore, HIV-positive patients are excluded from the study because of possible lethal side effects.
* Bulk disease (tumor volume > 70% of the target liver volume, or tumor nodules too numerous to count)
* Aspartic transaminase (AST) or alanine transaminase (ALT) > 5 times upper limit of normal (ULN)
* Bilirubin > 2 mg/dL
* Child-Pugh C Liver Cirrhosis
* Tumor volume > 50% combined with an albumin < 3 g/dL
* Complete occlusion of main portal vein causing portal hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hoffe, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-five participants were enrolled at Moffitt Cancer Center between 2010 and 2013.
Period: Overall Study
Arm/Group | Arterial Injection of 90-Y Microspheres
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Arterial Injection of 90-Y Microspheres
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 20
Age, Continuous [Median (Full Range); unit: years] | 76 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from enrollment to time of progression or death from any cause. Progression will be defined as progressive disease in the treated lobe. If progression is seen in a treated lobe, this will be considered a treatment failure. Progressive Disease (PD) according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST) Version 1.1.: At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: End of post treatment follow-up period of 20 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arterial Injection of 90-Y Microspheres
Number analyzed (Participants) | 25
months | 6 [4 to 12]

2. Secondary Outcome: Median Overall Survival (OS)
Description: OS is defined as the duration of time from enrollment to time of death from any cause.
Time Frame: Up to 36 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arterial Injection of 90-Y Microspheres
Number analyzed (Participants) | 25
months | 22 [10 to NA] — Upper limit not reached

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Tumor Response according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Complete Response (CR): Complete disappearance of all target and non-target lesions; no new lesions. Partial Response (PR): Applies only to patients with at least one measurable lesion; Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions; No unequivocal progression of non-measurable disease; No new lesions.
Time Frame: End of post treatment follow-up period of up to 20 months
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Arterial Injection of 90-Y Microspheres
Number analyzed (Participants) | 25
percentage of participants | 56

ADVERSE EVENTS:
Time Frame: 4 years, 5 months
Arm/Group | Arterial Injection of 90-Y Microspheres
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arterial Injection of 90-Y Microspheres (N=25)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Infections and infestations - Other, urosepsis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Blood bilirubin increased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arterial Injection of 90-Y Microspheres (N=25)
Fatigue (General disorders) | 23 (34)
Flu like symptoms (General disorders) | 7 (8)
Edema limbs (General disorders) | 5 (6)
Chills (General disorders) | 3 (4)
Pain (General disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 23 (37)
Alkaline phosphatase increased (Investigations) | 20 (27)
Aspartate aminotransferase increased (Investigations) | 7 (8)
Platelet count decreased (Investigations) | 6 (8)
Weight loss (Investigations) | 6 (6)
Blood bilirubin increased (Investigations) | 4 (6)
Alanine aminotransferase increased (Investigations) | 5 (6)
White blood cell decreased (Investigations) | 4 (5)
Activated partial thromboplastin time prolonged (Investigations) | 3 (4)
Creatinine increased (Investigations) | 3 (4)
INR increased (Investigations) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 20 (30)
Nausea (Gastrointestinal disorders) | 18 (28)
Dyspepsia (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 13 (16)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (12)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 15 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hot flashes (Vascular disorders) | 4 (5)
Hypertension (Vascular disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes